CLINICAL TRIAL: NCT01937312
Title: Additive Effect of Brinzolamide 1%/Brimonidine 0.2% Fixed Dose Combination as Adjunctive Therapy to a Prostaglandin Analogue
Brief Title: Effect of SIMBRINZA® Suspension as an Added Therapy to a Prostaglandin Analogue
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-13-020
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
Keywords: glaucoma; prostaglandin analogue; brinzolamide; brimonidine
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Glaucoma | interventions — brinzolamide; Brimonidine Tartrate; Prostaglandins, Synthetic; Travoprost; Bimatoprost; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIMBRINZA (Experimental): Brinzolamide 1%/brimonidine 0.2% ophthalmic suspension, 1 drop in each eye 3 times a day (8 AM, 3 PM, 10 PM), with prostaglandin analogue, 1 drop in each eye at bedtime, for 6 weeks
  Interventions: Drug: Brinzolamide 1%/brimonidine 0.2% ophthalmic suspension; Drug: Prostaglandin analogue
- Vehicle (Placebo Comparator): Inactive ingredients, 1 drop in each eye 3 times a day (8 AM, 3 PM, 10 PM), with prostaglandin analogue, 1 drop in each eye at bedtime, for 6 weeks
  Interventions: Drug: Vehicle; Drug: Prostaglandin analogue

INTERVENTIONS:
Drug: Brinzolamide 1%/brimonidine 0.2% ophthalmic suspension
  Other Names: SIMBRINZA® Suspension
  Arms: SIMBRINZA
Drug: Vehicle — Inactive ingredients used as a placebo comparator
  Arms: Vehicle
Drug: Prostaglandin analogue
  Other Names: TRAVATAN Z®; LUMIGAN®; XALATAN®

SUMMARY:
The purpose of this study is to demonstrate the additive effect of brinzolamide 1%/brimonidine 0.2% (SIMBRINZA® suspension) in subjects with either open angle glaucoma or ocular hypertension who are currently on a prostaglandin analogue (PGA) monotherapy.

DETAILED DESCRIPTION:
This study was divided into 2 sequential phases. The Screening/Eligibility Phase included one Screening Visit and two Eligibility Visits, during which subjects washed out of all other intraocular pressure (IOP)-lowering medications and dosed with TRAVATAN Z®, XALATAN®, or LUMIGAN®, 1 drop instilled in each eye once daily for 28 days. Subjects who met all inclusion/exclusion criteria were randomized at the second Eligibility Visit. The Treatment Phase consisted of two on-therapy visits (Week 2 and Week 6).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open angle glaucoma (including open-angle glaucoma with pseudoexfoliation or pigment dispersion) or ocular hypertension;
* Mean intraocular pressure (IOP) measurements in at least 1 eye (study eye) of ≥ 21 mmHg and <32 mmHg at 2 consecutive visits (Eligibility 1 and Eligibility 2);
* Previously prescribed TRAVATAN Z® 0.004%, XALATAN® 0.005%, or LUMIGAN® 0.01% monotherapy for at least 28 days prior to the Screening Visit;
* Able to understand and sign Informed Consent Document;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential who are pregnant, breastfeeding, or do not agree to use an adequate birth control method throughout the study;
* Any form of glaucoma other than open angle glaucoma or ocular hypertension;
* Severe central visual field loss;
* Chronic, recurrent, or severe inflammatory eye disease;
* Ocular trauma within the past 6 months;
* Ocular infection or ocular inflammation within the past 3 months;
* Best-corrected visual acuity score worse than approximately 20/80 Snellen;
* Eye surgery within the past 6 months;
* Any condition, including severe illness, which would make the subject unsuitable for the study in the opinion of the Investigator;
* Use of any additional topical or systemic ocular hypertensive medication during the study;
* Patients who, in the opinion of the Investigator, cannot discontinue all IOP-lowering ocular medication(s) per the appropriate washout schedule prior to Eligibility 1 Visit;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Burmaster, PhD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled from 30 investigative sites located in the US.
Pre-assignment Details: Of the 282 enrolled, 93 participants were exited from the study as screen failures prior to randomization. This reporting group includes all randomized participants (189). Note: One subject randomized to SIMBRINZA® Suspension was not exposed to investigational product.
Groups:
- SIMBRINZA; Vehicle: 1 drop in each eye 3 times a day (8 AM, 3 PM, 10 PM), with prostaglandin analogue, 1 drop in each eye at bedtime, for 6 weeks
Period: Overall Study
Arm/Group | SIMBRINZA | Vehicle
Started | 94 | 95
Treated | 93 | 95
Completed | 83 | 92
Not Completed | 11 | 3
Not completed — Adverse Event | 10 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal of subject prior to treatment | 1 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who received study medication and completed at least 1 scheduled on-therapy visit (intent-to-treat).
Groups:
- Total: Total of all reporting groups
Arm/Group | SIMBRINZA | Vehicle | Total
Number analyzed (Participants) | 88 | 94 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (9.4) | 64.7 (9.6) | 65.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 63 | 116
  Male | 35 | 31 | 66
Mean Diurnal Intraocular Pressure (IOP) at Baseline [Mean (Standard Deviation); unit: mmHg] — Diurnal IOP at Baseline was defined as the average of the four Baseline IOP measurements at timepoints 8 AM, 10 AM, 3 PM, and 5 PM. For each timepoint, the baseline IOP was defined as the average of the timepoint-matched IOP measurements at the Eligibility 1 and Eligibility 2 Visits.
  mmHg | 22.68 (2.123) | 22.39 (2.774) | 22.53 (2.478)

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal Intraocular Pressure (IOP) at Week 6
Description: Diurnal IOP was defined as the average of the four timepoints measured (8 AM, 10 AM, 3 PM, and 5 PM). IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters mercury (mmHg). One eye was chosen as the study eye and only data for the study eye were used for the analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Week 6
Population: This analysis population includes all subjects who received study medication and completed at least 1 scheduled on-therapy visit (intent-to-treat). Last observation carried forward (LOCF) was not utilized; therefore, results report subjects present at Week 6 with no imputation for missingness.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIMBRINZA | Vehicle
Number analyzed (Participants) | 83 | 92
mmHg | 17.01 (2.897) | 20.37 (3.914)

2. Secondary Outcome: Mean Diurnal IOP Change From Baseline to Week 6
Description: Baseline IOP was defined as the average of the timepoint-matched IOP measurements at Eligibility 1 and Eligibility 2 Visits. Diurnal IOP change was defined as the average of the four changes from baseline (timepoints 8 AM, 10 AM, 3 PM, and 5 PM). IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters mercury (mmHg). One eye was chosen as the study eye and only data for the study eye were used for the analysis. A more negative change from baseline indicates a greater improvement, i.e., a reduction of IOP.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIMBRINZA | Vehicle
Number analyzed (Participants) | 83 | 92
mmHg | -5.69 (2.571) | -1.99 (2.865)

3. Secondary Outcome: Mean Diurnal IOP Percentage Change From Baseline to Week 6
Description: Baseline IOP was defined as the average of the timepoint-matched IOP measurements at Eligibility 1 and Eligibility 2 Visits. Diurnal IOP Percentage Change was defined as the average of the four percent changes from baseline (timepoints 8 AM, 10 AM, 3 PM, and 5 PM). IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters mercury (mmHg). One eye was chosen as the study eye and only data for the study eye were used for the analysis. A more negative percent change from baseline indicates a greater amount of improvement, i.e., a reduction of IOP.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SIMBRINZA | Vehicle
Number analyzed (Participants) | 83 | 92
percent change | -24.88 (10.818) | -8.50 (12.396)

4. Secondary Outcome: Mean IOP at Week 6 for Each Time Point (8 AM, 10 AM, 3 PM, 5 PM)
Description: IOP was assessed using Goldmann applanation tonometry and reported in mmHg. One eye was chosen as the study eye and only data for the study eye were used for the analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIMBRINZA | Vehicle
Number analyzed (Participants) | 83 | 92
mmHg
  8 AM | 19.4 (3.53) | 21.4 (4.33)
  10 AM | 15.8 (3.54) | 20.2 (4.17)
  3 PM | 17.2 (3.15) | 19.9 (4.28)
  5 PM | 15.6 (3.14) | 19.9 (4.41)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study, Oct 2013-May 2014. Adverse events are reported as pre-treatment and treatment-emergent. The treatment-emergent analysis set included all subjects exposed to investigational product.
Description: An AE was defined as any untoward medical occurrence in a subject who was administered a study medication, regardless of whether or not the event had a causal relationship with the medication. All AEs were obtained as solicited and spontaneous comments from the subjects, and as observations by the Investigator, as outlined in the study protocol.
Groups:
- Pre-Treatment: Prostaglandin analogue, 1 drop in each eye at bedtime for a 4-week run-in period
Arm/Group | Pre-Treatment | SIMBRINZA | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/282 | 1/93 | 0/95
Other Adverse Events (participants affected / at risk) | 2/282 | 16/93 | 8/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Treatment (N=282) | SIMBRINZA (N=93) | Vehicle (N=95)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Treatment (N=282) | SIMBRINZA (N=93) | Vehicle (N=95)
Vision Blurred (Eye disorders) | 0 | 9 | 6
Eye irritation (Eye disorders) | 1 | 6 | 1
Eye Pruritus (Eye disorders) | 0 | 6 | 0
Ocular hyperaemia (Eye disorders) | 2 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.